CLINICAL TRIAL: NCT02865993
Title: May Betadine Improve Cesarean Section Outcomes?
Brief Title: Betadine Irrigation in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Roberto Angioli, Full Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BetadineCS0405
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Infection; Cesarean Section
Keywords: cesarean section; cesarean section complications; betadine irrigation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betadine Group (Other): Patients intra-operatively received intraperitoneal irrigation prior to abdominal closure with low molecular weight povidone-iodine solution ('Betadine LMW') (PVP-I LMW) diluted 50:50 with normal saline.
  Interventions: Other: betadine group
- No Betadine Group (Other): Patients intra-operatively received intraperitoneal irrigation prior to abdominal closure with only normal saline solution.
  Interventions: Other: no betadine group

INTERVENTIONS:
Other: betadine group — Patients intra-operatively received intraperitoneal irrigation prior to abdominal closure with low molecular weight povidone-iodine solution ('Betadine LMW') (PVP-I LMW) diluted 50:50 with normal saline.
  Arms: Betadine Group
Other: no betadine group — Patients intra-operatively received intraperitoneal irrigation prior to abdominal closure with only normal saline solution.
  Arms: No Betadine Group

SUMMARY:
The purpose of this study was to evaluate, for the first time in Literature, the effects of betadine washing versus normal saline washing after uterine closure in women undergoing cesarean section (CS) at ≥36 gestational weeks in terms of post CS infections, complication, fever and pain.

DETAILED DESCRIPTION:
This was a single-centre randomized controlled trial performed at Department of Obstetrics and Gynecology of San Camillo Hospital of Rome. The protocol was approved by the Internal Review Board. All women having a cesarean section (CS) were eligible for recruitment unless there was suspected or known allergy to iodine. The study was widely publicized around obstetrics unit and all women were provided antenatally with a brief statement regarding the study. The study was presented to women as part of hospital initiative to reduce postoperative infections and to improve postoperative recovery. Consent was obtained from all women at the time of consenting for CS.

Background was recorded for each patient: maternal age, gestational week at delivery, BMI, and pregnancy complication; plural fetal pregnancies, premature rupture of membranes, placenta previa and pre-eclampsia. The investigators recorded the type of cesarean procedure, elective (scheduled operations) or urgent (patients in labor and maternal or fetal emergent indication), mean surgical time to perform CS.

In Literature, povidone-iodine irrigation has been demonstrated to be a simple and inexpensive solution with the potential to prevent surgical site infection , which can also reduce the incidence of intra-abdominal infectious complications when used as an intraperitoneal irrigant in patients undergoing bacterially-contaminated surgical procedures, i.e. orthopedic, general surgery, oncologic surgery. Therefore, the investigators aimed to test its use in CS.

Patients were intra-operatively randomized to receive intraperitoneal irrigation prior to abdominal closure with low molecular weight povidone-iodine solution ('Betadine LMW') (PVP-I LMW) diluted 50:50 with normal saline or with only normal saline solution. Randomization to 'Betadine' or 'no Betadine' group was performed using sequentially numbered sealed opaque envelopes that contained the allocation. The allocation was prepared using computer generated list of random numbers using a variable block of 10 and performed by a staff members, part of the clinical team. After all layers were sutured and just prior to starting skin closure, the envelope with the allocation was opened by one of the theatre nurse.

All CS were generally performed under spinal anesthesia by the specialist obstetricians, credentialed trainee registrars or by juniors in the presence of a specialist obstetrician using the modified Misgav Ladach surgical technique.

An abdominal opening was made through a straight transverse incision, which was placed 3-4 cm above the symphysis. The subcutaneous tissue was left untouched apart from the midline. The rectus sheath was separated along its fibers and the rectus muscles separated by pulling. Stretching with index fingers opened the peritoneum and the uterus was opened with an index finger. The hole was enlarged between the index finger of one hand and the thumb of the other.

Single-layer closure of the uterine incision was performed as follows: a holding Vicryl-0 was placed in the left corner to stabilize and define the demarcation of the suture line. A continuous non-locking stitch beginning at the right corner was used, closing the whole thickness of the uterine wall, excluding the decidual layer, in a cranial/caudal position. Additional single sutures were added for hemostasis if required. Routinely exteriorization of the uterus was not performed. The visceral and parietal peritoneal layers were left open and the rectus muscle was not stitched. The rectus sheath was stitched with a continuous non-locking Vicryl-0 and the subdermal space was closed in all patients. All patients had preoperative exams not longer than 4 weeks prior the CS and received prophylactic intravenous antibiotics (amoxicillin 2 g and metronidazole 1 g) preoperatively to reduce the rate of wound infection. In addition, all patients received oxytocin intravenous during CS and 20 IU was administered by an intravenous drip running post surgical procedure. All patients were encouraged to start breastfeeding during early postoperative care, supported by a midwife and by a nurse specialized in newborn care after admission to the maternity ward.

Post CS infections included:

* Postpartum endometritis: defined as a clinical diagnosis, usually involving fever, uterine fundal tenderness, or purulent lochia requiring antibiotic therapy.
* Postoperative wound infection: defined as erythema, tenderness, purulent drainage from the incision site, with or without fever, requiring antibiotic therapy.
* Postoperative fever: defined as greater than 38 degrees C or 100.4 degrees F.
* Postoperative wound seroma or hematoma: defined as collection of serous fluid or blood/clot in the subcutaneous area of the incision.
* Composite wound complications: defined as the presence of any one of the following: wound infection, seroma, hematoma, separation.

Patients were examined during daily rounds whilst in hospital about intestinal recanalization, postoperative mobilization, postoperative 24h post CS pain and wounds. Preoperative and postoperative exams, presence of fever or any symptoms have been accurately registered.

After discharge from the hospital, the women were sent a letter with addressed return envelope to report any post CS problems at four weeks after surgery as part of hospital surveillance policy. Charts of all women readmitted for any reason were reviewed. Differences between 'Betadine' and 'no Betadine' groups were assessed using chi square for categorical data test. Fisher's exact test was used where there were 5 or fewer counts within a category and t-test for continuous data. Relative risk (RR) and the corresponding 95% confidence interval (CI) were calculated. A P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50 years
* planned or urgent cesarean section (CS)
* gestational age > 36 weeks
* written informed consent

Exclusion criteria:

* suspected or known allergy to iodine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative infections | up to 20 days after cesarean section
  postoperative infections expressed in number of patients with postoperative infections, such as endometritis or wood infections up to 20 days after cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Angioli, Professor, Study Director — Campus Bio-Medico University
Locations (1):
- campus bio-medico of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided